CLINICAL TRIAL: NCT03999073
Title: Carotid Atherosclerosis in Patients With Aortic Coarctation
Acronym: CoA
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Joanna Hlebowicz, MD, Associated Professor, Skane University Hospital
Other Study IDs: 2017/260
Record Dates: First submitted 2019-06-21; First posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Atherosclerosis; Aortic Coarctation
MeSH Terms: conditions — Atherosclerosis; Aortic Coarctation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with coarctation
  Interventions: Other: Ultrasound measurement
- Controls
  Interventions: Other: Ultrasound measurement

INTERVENTIONS:
Other: Ultrasound measurement — Ultrasound measurement

SUMMARY:
Despite aortic coarctation (CoA) repair these patients have cardiovascular complications and coronary artery disease is the most common cause of death.

DETAILED DESCRIPTION:
The aim with this study was to measure intima-media thickness (IMT) and plaques in arteries compared to cardiovascular markers in controls and patients with CoA.

ELIGIBILITY:
Inclusion Criteria:

* sex and age-matched controls

Exclusion Criteria:

* acute and chronic inflammation disease, underlying malignancies and diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — sex and age-matched controls
Study Population: Patients with aortic coarctation
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Intima-media thickness | Intima-media thickness will be measured at one time point namely at inclusion. Data will be reported when study is completed, an average of 2 year.
  Measurement in mm

SECONDARY OUTCOMES:
Cardiovascular markers | Blood samples will be taken at one time point namely at inclusion. Then biomarkers will be analysed when study is completed. Data will be reported when study is completed, an average of 2 year.
  A multiplex platform to analyze circulating blood levels biomarkers was used.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hlebowicz J, Holm J, Lindstedt S, Goncalves I, Nilsson J. Carotid atherosclerosis, changes in tissue remodeling and repair in patients with aortic coarctation. Atherosclerosis. 2021 Oct;335:47-52. doi: 10.1016/j.atherosclerosis.2021.09.016. Epub 2021 Sep 21. PMID 34564048